CLINICAL TRIAL: NCT00233142
Title: Expressive Writing: Complementary Treatment for Diabetes
Brief Title: Expressive Writing for Reducing Stress and Diabetic Symptoms in Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT002477 (NIH); R01AT002477 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-10-05 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes Mellitus; Stress; Depression
Keywords: Diabetes; Emotions; Blood glucose; Expressive Writing
MeSH Terms: conditions — Diabetes Mellitus; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Expressive writing (Experimental): Expressive writing
  Interventions: Behavioral: Expressive writing
- Neutral writing (Sham Comparator): Non-expressive writing
  Interventions: Behavioral: Neutral writing

INTERVENTIONS:
Behavioral: Expressive writing — Writing as therapeutic intervention
  Arms: Expressive writing
Behavioral: Neutral writing — Non-expressive writing
  Arms: Neutral writing

SUMMARY:
This study will determine whether the psychological benefits of expressive writing extend to diabetic patients, how long the benefits will last, and whether additional expressive writing "booster" sessions will lead to greater and more sustained improvement in diabetes symptoms and well-being.

DETAILED DESCRIPTION:
Diabetes is one of the leading causes of blindness, kidney failure, and nontraumatic lower extremity amputation in the United States. Conditions such as stress and depression have been shown to worsen diabetic symptoms. Data indicate that expressive writing (an activity during which individuals deal with stressful experiences by writing about them on paper) has beneficial effects on psychological and physiological outcomes. This study will determine whether diabetes patients can benefit from expressive writing. This study will also determine the duration of the benefits and the effectiveness of booster sessions in improving their diabetic symptoms.

Participants will be randomly assigned to engage in expressive writing or neutral writing for 18 months. Participants in the expressive writing group will write about traumatic or stressful events; participants in the neutral writing group will write about neutral topics that do not affect them emotionally. Some participants in the expressive writing group will receive an additional 4 months of booster sessions of expressive writing. All participants will undergo interviews, blood collection, physical exams and complete clinical scales on their disease status, quality of life, and psychological well-being; these assessments will occur at study entry, every 4 months during the study, and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus made after age 24

Exclusion Criteria:

* Diabetes-related emergency room visit within 3 months prior to study entry
* Use of psychiatric medication within 3 months prior to study entry
* Visual or manual limitations that preclude reading and writing
* Use of insulin within the first year of diabetes diagnosis
* Pregnancy or plan to become pregnant

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2005-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1C (indicator of blood glucose) | baseline, 4 months, 8 months, 12 months, and 16 months

SECONDARY OUTCOMES:
Diabetes symptoms | baseline, 4 months, 8 months, 12 months, and 16 months
stress levels | baseline, 4 months, 8 months, 12 months, and 16 months
depression | baseline, 4 months, 8 months, 12 months, and 16 months
cognitive function | baseline, 4 months, 8 months, 12 months, and 16 months
quality of life | baseline, 4 months, 8 months, 12 months, and 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M. Smyth, PhD, Principal Investigator — Syracuse University
Locations (4):
- United States (4):
  - State University of New York Medical University, Syracuse, New York
  - Syracuse University, Syracuse, New York
  - Pennsylvania State University, University Park, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee